CLINICAL TRIAL: NCT00803712
Title: Randomized Trial to Evaluate the Efficacy and Safety of Cinacalcet Treatment in Combination With Low Dose Vitamin D for the Treatment of Subjects With Secondary Hyperparathyroidism (SHPT) Recently Initiating Hemodialysis
Brief Title: 20070360 Incident Dialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070360
Record Dates: First submitted 2008-11-26; First posted 2008-12-05 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Chronic Kidney Disease; Secondary Hyperparathyroidism
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — Cinacalcet; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cinacalcet Group (Experimental): Cinacalcet plus low dose active Vitamin D (if prescribed)
  Interventions: Drug: Cinacalcet
- Control Group (Active Comparator): Flexible active vitamin D dosing
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Cinacalcet — Cinacalcet is a calcimimetic agent, which is synthesized as a hydrochloride salt.
  Other Names: Sensipar/Mimpara
  Arms: Cinacalcet Group
Drug: Vitamin D — Titration of active Vitamin D in accordance with treatment practice guidelines in order to treat Secondary Hyperparathyroidism.
  Other Names: Active Vitamin D
  Arms: Control Group

SUMMARY:
Randomized Trial to Evaluate the Efficacy and Safety of Cinacalcet Treatment in Combination with Low Dose Vitamin D for the Treatment of Subjects with Secondary Hyperparathyroidism (SHPT) Recently Initiating Hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to 18 years of age on hemodialysis for > 3 and less than or equal to 12 months prior to enrollment into the study
* Mean of 2 PTH determinations during the screening period (drawn at least 2 days apart) > 300 pg/mL (31.8 pmol/L); or biPTH > 160 pg/mL (17.0 pmol/L)
* Mean of 2 corrected serum calcium determinations drawn on the same day as the PTH determinations greater than or equal to 8.4 mg/dL (2.1 mmol/L)
* Subject will be able to complete the study, to the best of his/her knowledge
* Before any study-specific procedure, the appropriate written informed consent must be obtained

Exclusion Criteria:

* Mean of 2 PTH determinations during the screening period (drawn at least 2 days apart) > 800 pg/mL (84.9 pmol/L); or biPTH > 430 pg/mL (45.6 pmol/L) AND receiving vitamin D on entering screening
* Parathyroidectomy (partial or full) less than or equal to 6 months before entering screening
* Anticipated parathyroidectomy (partial or full) within 6 months after randomization
* Have a scheduled date for kidney transplant surgery
* Received cinacalcet since initiating hemodialysis
* Have received vitamin D therapy for less than 30 days before entering screening or required a change in prescribed vitamin D brand or dose within 30 days before entering screening. If subjects are not receiving vitamin D therapy, they must remain free of vitamin D therapy for the 30 days before entering screening
* Subject is pregnant (eg, positive HCG test) or is breast-feeding
* Refusal to use highly effective contraceptive measures (as determined by the investigator) throughout the study (screening and post enrollment)
* Current gastrointestinal disorder that may be associated with impaired absorption of orally administered medications or an inability to swallow tablets
* Known sensitivity, intolerance, or other adverse response to cinacalcet which would prevent on-study treatment compliance
* Have an unstable medical condition within 30 days before screening, or otherwise unstable in the judgment of the investigator
* Subject is currently enrolled in, or fewer than 30 days prior to entering screening have passed since subject received other investigational agent(s) (devices or drug).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2010-12-09 (Actual); Study Completion 2011-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Rodriguez M, Urena-Torres P, Petavy F, Cooper K, Farouk M, Goodman WG. Calcium-mediated parathyroid hormone suppression to assess progression of secondary hyperparathyroidism during treatment among incident dialysis patients. J Clin Endocrinol Metab. 2013 Feb;98(2):618-25. doi: 10.1210/jc.2012-3246. Epub 2013 Jan 30. PMID 23365129
- [Background] Urena-Torres P, Bridges I, Christiano C, Cournoyer SH, Cooper K, Farouk M, Kopyt NP, Rodriguez M, Zehnder D, Covic A. Efficacy of cinacalcet with low-dose vitamin D in incident haemodialysis subjects with secondary hyperparathyroidism. Nephrol Dial Transplant. 2013 May;28(5):1241-54. doi: 10.1093/ndt/gfs568. Epub 2013 Jan 16. PMID 23328710
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant was enrolled on 19 February 2009 and last participant completed the study on 5 July 2011. 313 participants were enrolled from 82 study centers in US, Europe, Canada, Australia and Russia.
Pre-assignment Details: Once participants were determined to be eligible for the study, they entered a pre-randomization wash-out phase of 4 weeks (if receiving vitamin D at the time of enrollment). Four enrolled participants did not complete the pre-randomization wash-out phase and were not randomized into the study.
Groups:
- Cinacalcet: cinacalcet in combination with low-dose active vitamin D (if prescribed)
- Control Group: Flexible active vitamin D dosing (if prescribed) per standard treatment guidelines.
Period: Overall Study
Arm/Group | Cinacalcet | Control Group
Started | 154 (154 participants were randomized to the cinacalcet group) | 155 (155 participants were randomized to the control group)
Full Analysis Set | 153 (153 participants randomized and had at least one PTH concentration available after study day 1.) | 151 (151 participants randomized and had at least one PTH concentration available after study day 1.)
Safety Analysis Set | 155 (Rz'ed to cinacalcet and received at least 1 dose, or to control but received cinacalcet throughout) | 154 (Randomized to the control group)
Completed | 118 (118 participants randomized to the cinacalcet group completed the study) | 128 (128 participants randomized to the control group completed the study)
Not Completed | 36 | 27
Not completed — Noncompliance | 3 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Death | 8 | 7
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — "Other" in electronic Case Report Form | 0 | 1
Not completed — Protocol criteria (other) | 0 | 2
Not completed — Protocol criteria (renal transplant) | 12 | 8
Not completed — Administrative decision | 2 | 3
Not completed — Protocol criteria (parathyroidectomy) | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cinacalcet | Control Group | Total
Number analyzed (Participants) | 153 | 151 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (13.6) | 57.0 (14.6) | 57.4 (14.1)
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 105 | 99 | 204
  >=65 years | 48 | 52 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 56 | 126
  Male | 83 | 95 | 178
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 120 | 111 | 231
  Black or African American | 28 | 31 | 59
  Hispanic or Latino | 1 | 1 | 2
  Asian | 3 | 5 | 8
  Aborigine | 0 | 1 | 1
  Other | 1 | 2 | 3
Active Vitamin D Use [Number; unit: participants] — Active Vitamin D use at baseline
  participants
    Active Vitamin D use | 74 | 72 | 146
    No active Vitamin D use | 79 | 79 | 158
iPTH [Mean (Standard Deviation); unit: pg/mL] — iPTH value at baseline
  pg/mL | 559.2 (338.2) | 511.6 (253.6) | 535.5 (299.6)
Corrected Serum Calcium [Mean (Standard Deviation); unit: mg/dL] — Corrected serum calcium at baseline
  mg/dL | 9.30 (0.69) | 9.14 (0.49) | 9.22 (0.60)
Serum Phosphorus [Mean (Standard Deviation); unit: mg/dL] — serum phosphorus at baseline
  mg/dL | 5.55 (1.70) | 5.49 (1.60) | 5.52 (1.65)
Albumin [Mean (Standard Deviation); unit: g/dL] — Albumin at baseline
  g/dL | 3.93 (0.39) | 3.89 (0.40) | 3.91 (0.39)
Dialysis Vintage [Mean (Standard Deviation); unit: months] — Time since dialysis started
  months | 7.29 (2.54) | 7.02 (2.78) | 7.16 (2.66)

OUTCOME MEASURES:

1. Primary Outcome: Achievement of a ≥ 30% Reduction in Mean PTH From Baseline to During the Efficacy Assessment Phase at Month 6 (Weeks 22 to 26)
Description: All available measurements from the efficacy assessment phase (EAP) at month 6 were used in the calculation of the mean over the period. For participants with no measurements taken during the EAP, the mean of the last 2 measurements available after Day 1 were carried forward. If there was only 1 value available, this single value was carried forward to the EAP.
Time Frame: Weeks 22-26
Population: Analysis based on the full analysis set, including all participants who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for participants without an iPTH value during weeks 22-26
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders defined as >= 30% reduction in Mean PTH | 96 | 58
  Non responders | 57 | 93
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Hypothesis to be tested: the proportion of participants achieving the specified PTH target of ≥ 30% reduction in PTH from baseline will be greater in the cinacalcet plus low dose active vitamin D group than in the control group during the efficacy assessment phase at month 6 (weeks 22 to 26); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Achievement of a Mean PTH <= 300 pg/mL During the Efficacy Assessment Phase at Month 6 (Weeks 22 to 26)
Description: All available measurements from the efficacy assessment phase (EAP) at month 6 were used in the calculation of the mean over the period. For subjects with no measurements taken during the EAP, the mean of the last 2 measurements available after Day 1 were carried forward. If there was only 1 value available, this single value was carried forward to the EAP.
Time Frame: Weeks 22-26
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without an iPTH value during weeks 22-26
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders defined as a mean PTH <= 300 pg/mL | 87 | 53
  Non responders | 66 | 98
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is presented, adjusted using the Dubey and Armitage-Parmer method

3. Secondary Outcome: Achievement of a ≥ 30% Reduction in Mean PTH From Baseline to During the Efficacy Assessment Phase at Month 12 (Weeks 48 to 52)
Description: All available measurements from the efficacy assessment phase (EAP) at month 12 were used in the calculation of the mean over the period. For subjects with no measurements taken during the EAP, the mean of the last 2 measurements available after Day 1 were carried forward. If there was only 1 value available, this single value was carried forward to the EAP.
Time Frame: Weeks 48-52
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without an iPTH value during weeks 48-52
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders defined as >= 30% reduction in mean PTH | 97 | 72
  Non responders | 56 | 79
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.0139, Cochran-Mantel-Haenszel — Adjusted p-value is presented. P-value is adjusted using Dubey and Armitage-Parmer method of adjusting for multiple comparisons

4. Secondary Outcome: Achievement of a Mean PTH <= 300 pg/mL During the Efficacy Assessment Phase at Month 12 (Weeks 48 to 52)
Description: as for outcome 3
Time Frame: Weeks 48-52
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders defined as a mean PTH <= 300 pg/mL | 80 | 67
  Non responders | 73 | 84
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.2386, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is presented, adjusted using the Dubey and Armitage-Parmer method

5. Secondary Outcome: Achievement of a Mean Corrected Serum Calcium < 10.2 mg/dL During the Efficacy Assessment Phase at Month 6 (Weeks 22 to 26)
Description: as for outcome 2
Time Frame: Weeks 22-26
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without a corrected serum calcium value during weeks 22-26
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders, a mean corrected calcium < 10.2 mg/dL | 151 | 144
  Non responders | 2 | 7
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.0875, Cochran-Mantel-Haenszel

6. Secondary Outcome: Achievement of a Mean Corrected Serum Calcium < 10.2 mg/dL During the Efficacy Assessment Phase at Month 12 (Weeks 48 to 52)
Description: as for outcome 3
Time Frame: Weeks 48-52
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without a corrected serum calcium value during weeks 48-52
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders, a mean corrected calcium < 10.2 mg/dL | 146 | 141
  Non responders | 7 | 10
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.4304, Cochran-Mantel-Haenszel

7. Secondary Outcome: Achievement of a Mean Serum Phosphorus < 5.5 mg/dL During the Efficacy Assessment Phase at Month 6 (Weeks 22 to 26)
Description: as for outcome 2
Time Frame: Weeks 22-26
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without a serum phosphorus value during weeks 22-26
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders, a mean phosphorus < 5.5 mg/dL | 100 | 85
  Non responders | 53 | 66
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.0910, Cochran-Mantel-Haenszel

8. Secondary Outcome: Achievement of a Mean Serum Phosphorus < 5.5 mg/dL During the Efficacy Assessment Phase at Month 12 (Weeks 48 to 52)
Description: as for outcome 3
Time Frame: Weeks 48-52
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without a serum phosphorus value during weeks 48-52
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders, a mean serum phosphorus < 5.5 mg/dL | 81 | 80
  Non responders | 72 | 71
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.9520, Cochran-Mantel-Haenszel

9. Secondary Outcome: Achievement of a >= 30% Reduction in Mean iPTH From Baseline to During Both Efficacy Assessment Phases at Month 6 (Weeks 22 to 26) and Month 12 (Weeks 48 to 52)
Description: All available measurements from the efficacy assessment phases were used in the calculation of the mean over the period. For subjects with no measurements taken during an EAP, the mean of the last 2 measurements available after Day 1 were carried forward. If there was only 1 value available, this single value was carried forward to the EAP.
Time Frame: Weeks 22-26 and Weeks 48-52
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without an iPTH value during the efficacy assessment phases
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders, a >= 30% reduction in mean iPTH | 74 | 42
  Non responders | 79 | 109
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel

10. Secondary Outcome: Achievement of a Mean iPTH <=300 pg/mL During Both Efficacy Assessment Phases at Month 6 (Weeks 22 to 26) and Month 12 (Weeks 48 to 52)
Description: as for outcome 9
Time Frame: Weeks 22-26 and Weeks 48-52
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders, a mean iPTH <= 300 pg/mL | 54 | 39
  Non responders | 99 | 112
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.0611, Cochran-Mantel-Haenszel

11. Secondary Outcome: Achievement of a Mean Corrected Serum Calcium < 10.2 mg/dL During Both Efficacy Assessment Phases at Month 6 (Weeks 22 to 26) and Month 12 (Weeks 48 to 52)
Description: as for outcome 9
Time Frame: Weeks 22-26 and Weeks 48-52
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without a corrected serum calcium value during the efficacy assessment phases
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders, a mean corrected calcium < 10.2 mg/dL | 145 | 139
  Non responders | 8 | 12
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.3298, Cochran-Mantel-Haenszel

12. Secondary Outcome: Achievement of a Mean Serum Phosphorus < 5.5 mg/dL During Both Efficacy Assessment Phases at Month 6 (Weeks 22 to 26) and Month 12 (Weeks 48 to 52)
Description: as for outcome 9
Time Frame: Weeks 22-26 and Weeks 48-52
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without a serum phosphorus value during the efficacy assessment phases
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
participants
  Responders, a mean serum phosphorus < 5.5 mg/dL | 71 | 64
  Non responders | 82 | 87
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.4436, Cochran-Mantel-Haenszel

13. Secondary Outcome: Summary of iPTH (pg/mL) at Month 6 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 22-26
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without an iPTH value during the efficacy assessment phase
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
pg/mL | 291.15 [264.24 to 320.81] | 402.11 [364.51 to 443.59]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis was adjusted for randomization strata. Due to distributional properties of the data, analysis was performed on log-transformed data

14. Secondary Outcome: Summary of Percent Change From Baseline in iPTH (pg/mL) at Month 6 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 22-26
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
percent change | -34.62 [-41.32 to -27.93] | -9.69 [-16.47 to -2.91]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis was adjusted for randomization strata

15. Secondary Outcome: Summary of iPTH (pg/mL) at Month 12 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 48-52
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
pg/mL | 293.95 [262.92 to 328.64] | 364.79 [325.84 to 408.40]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.0040, ANCOVA; [statistical method as in outcome 13, analysis 1]

16. Secondary Outcome: Summary of Percent Change From Baseline in iPTH (pg/mL) at Month 12 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 48-52
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
percent change | -34.15 [-41.96 to -26.33] | -12.41 [-20.32 to -4.49]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis was adjusted for randomization strata

17. Secondary Outcome: Summary of Corrected Serum Calcium (mg/dL) at Month 6 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 22-26
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without a corrected serum calcium value during the efficacy assessment phase
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
mg/dL | 8.66 [8.56 to 8.76] | 9.30 [9.20 to 9.40]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis was adjusted for randomization strata and baseline corrected serum calcium

18. Secondary Outcome: Summary of Percent Change From Baseline in Corrected Serum Calcium at Month 6 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 22-26
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
percent change | -5.68 [-6.73 to -4.63] | 1.05 [-0.01 to 2.12]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis was adjusted for randomization strata and baseline corrected serum calcium

19. Secondary Outcome: Summary of Corrected Serum Calcium (mg/dL) at Month 12 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 48-52
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
mg/dL | 8.95 [8.85 to 9.06] | 9.42 [9.32 to 9.53]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis was adjusted for randomization strata and baseline corrected serum calcium

20. Secondary Outcome: Summary of Percent Change From Baseline in Corrected Serum Calcium at Month 12 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 48-52
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
percent change | -2.62 [-3.72 to -1.51] | 2.37 [1.25 to 3.49]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis was adjusted for randomization strata and baseline corrected serum calcium

21. Secondary Outcome: Summary of Serum Phosphorus (mg/dL) at Month 6 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 22-26
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started. Last observation carried forward was used for subjects without a serum phosphorus value during the efficacy assessment phase
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
mg/dL | 5.11 [4.88 to 5.34] | 5.52 [5.29 to 5.75]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.0085, ANCOVA; Analysis was adjusted for randomization strata and baseline serum phosphorus

22. Secondary Outcome: Summary of Percent Change From Baseline in Serum Phosphorus at Month 6 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 22-26
Population: as for outcome 21
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
percent change | -1.79 [-6.51 to 2.93] | 3.94 [-0.87 to 8.75]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.0710, ANCOVA; Analysis was adjusted for randomization strata and baseline serum phosphorus

23. Secondary Outcome: Summary of Serum Phosphorus (mg/dL) at Month 12 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 48-52
Population: as for outcome 21
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
mg/dL | 5.37 [5.12 to 5.62] | 5.53 [5.27 to 5.78]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.3546, ANCOVA; Analysis was adjusted for randomization strata and baseline serum phosphorus

24. Secondary Outcome: Summary of Percent Change From Baseline in Serum Phosphorus at Month 12 Efficacy Assessment Phase
Description: as for outcome 9
Time Frame: Weeks 48-52
Population: as for outcome 21
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 153 | 151
percent change | 3.21 [-1.71 to 8.14] | 4.26 [-0.76 to 9.28]
Statistical Analysis 1: Comparison: Cinacalcet vs Control Group; Test type: Superiority or Other; p = 0.7518, ANCOVA; Analysis was adjusted for randomization strata and baseline serum phosphorus

25. Secondary Outcome: Subject Incidence of Hypercalcemia During the Efficacy Assessment Phase at Month 6
Description: Hypercalcemia is defined as at least one corrected serum calcium value >= 10.2 mg/dL
Time Frame: Weeks 22-26
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started, and also had at least one corrected serum calcium value during the time period of interest.
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 136 | 143
participants | 11 | 22

26. Secondary Outcome: Subject Incidence of Hypercalcemia During the Maintenance Phase
Description: Hypercalcemia is defined as at least one corrected serum calcium value >= 10.2 mg/dL
Time Frame: Weeks 26-48
Population: as for outcome 25
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 133 | 136
participants | 16 | 25

27. Secondary Outcome: Subject Incidence of Hypercalcemia During the Efficacy Assessment Phase at Month 12
Description: Hypercalcemia is defined as at least one corrected serum calcium value >= 10.2 mg/dL
Time Frame: Weeks 48-52
Population: as for outcome 25
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 119 | 128
participants | 15 | 21

28. Secondary Outcome: Subject Incidence of Hyperphosphatemia During the Efficacy Assessment Phase at Month 6
Description: Hyperphosphatemia is defined as at least one serum phosphorus value >= 5.5 mg/dL
Time Frame: Weeks 22-26
Population: Analysis based on the full analysis set, including all subjects who were randomized into the study and had at least one iPTH value available after the day study treatment started, and also had at least one serum phosphorus value during the time period of interest.
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 136 | 143
participants | 71 | 93

29. Secondary Outcome: Subject Incidence of Hyperphosphatemia During the Maintenance Phase
Description: Hyperphosphatemia is defined as at least one serum phosphorus value >= 5.5 mg/dL
Time Frame: Weeks 26-48
Population: as for outcome 28
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 133 | 138
participants | 71 | 87

30. Secondary Outcome: Subject Incidence of Hyperphosphatemia During the Efficacy Assessment Phase at Month 12
Description: Hyperphosphatemia is defined as at least one serum phosphorus value >= 5.5 mg/dL
Time Frame: Weeks 48-52
Population: as for outcome 28
Measure: Number; unit: participants
Arm/Group | Cinacalcet | Control Group
Number analyzed (Participants) | 119 | 128
participants | 74 | 83

ADVERSE EVENTS:
Time Frame: 56 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events. One patient randomized to the control group received cinacalcet throughout the study and is summarized in the cinacalcet arm for adverse events.
Arm/Group | Cinacalcet | Control Group
Serious Adverse Events (participants affected / at risk) | 72/155 | 52/154
Other Adverse Events (participants affected / at risk) | 107/155 | 87/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=155) | Control Group (N=154)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 5 | 1
Angina unstable (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 4
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 4
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Pericarditis uraemic (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 0 | 2
Catheter site discharge (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 3 | 3
Chills (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Hernia obstructive (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Nodule (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 5 | 1
Cellulitis gangrenous (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2
Groin infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 3
Localised infection (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 1 | 3
Postoperative wound infection (Infections and infestations) | 1 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 5 | 3
Septic embolus (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 4 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 7 | 3
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Chemical burn of skin (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 2 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Apraxia (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Convulsion (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Hemianopia (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Transverse sinus thrombosis (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Renal cyst ruptured (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypertensive crisis (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 3 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Poor peripheral circulation (Vascular disorders) | 0 | 1
Steal syndrome (Vascular disorders) | 2 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Venous stenosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=155) | Control Group (N=154)
Abdominal pain (Gastrointestinal disorders) | 4 | 8
Constipation (Gastrointestinal disorders) | 10 | 7
Diarrhoea (Gastrointestinal disorders) | 25 | 18
Nausea (Gastrointestinal disorders) | 30 | 15
Vomiting (Gastrointestinal disorders) | 26 | 13
Pyrexia (General disorders) | 8 | 12
Urinary tract infection (Infections and infestations) | 9 | 5
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 8 | 14
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 7 | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 8 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 25 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 8
Headache (Nervous system disorders) | 8 | 12
Insomnia (Psychiatric disorders) | 11 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 10
Hypertension (Vascular disorders) | 10 | 11
Hypotension (Vascular disorders) | 6 | 8

LIMITATIONS AND CAVEATS:
This was an open-label study and neither investigators nor subjects were blinded to treatment modality. Cinacalcet was dosed by forced titration. Active vitamin D administration was at the discretion of the investigator in each treatment arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.